CLINICAL TRIAL: NCT00584896
Title: A Phase 3 Clinical Trial to Assess Perfusion and Obstruction Identified by Non-Invasive Technology Using PB127 Ultrasound Contrast Agent in Patients With Suspected Obstructive Coronary Artery Disease II
Brief Title: Safety and Efficacy Study of PB127 Ultrasound Contrast Agent for Diagnosis of Coronary Artery Disease
Acronym: POINT II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued PB127 development program for business reasons
Sponsor: Point Biomedical (Industry)
Responsible Party: Tom Ottoboni, PhD/Chief Operating Officer, POINT Biomedical Corp.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127-014
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
Keywords: heart disease; coronary artery disease; echocardiogram; ultrasound; angiogram; SPECT; chest pain; perfusion
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PB127 for Injectable Suspension — 0.062 mg/kg continuous IV infusion (100-250 mL/hr) during echocardiography, not to exceed 60 minutes infusion, single dose.
  Other Names: CARDIOshpere®

SUMMARY:
The purpose of this study is to determine if the use of PB127 with cardiac ultrasound assists in the diagnosis or exclusion of coronary artery disease.

ELIGIBILITY:
1. 18 years old or older and able to provide written informed consent;
2. All subjects must be scheduled for or have undergone SPECT within 28 days prior to or following Study Day 1
3. Subjects with very low/low pre-test probability of coronary artery disease must consent to participate in the extension trial 127-014-A
4. Subjects with very low/low pre-test probability of coronary artery disease must not have a current diagnosis of obstructive CAD on angiogram or prior MI
5. Subjects with very low/low pre-test probability of coronary artery disease with a current diagnosis of obstructive CAD on angiogram or prior MI may be enrolled into Stratum 2
6. Subjects with intermediate or high pre-test probability of coronary artery disease must be scheduled for coronary angiography within the 28 days following Study Day 1
7. Sinus rhythm at the time of the study procedure
8. Adequate visualization of myocardial segments
9. Appropriate candidate for stress testing according to ACC/AHA Guidelines for Exercise Testing

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Known hypersensitivity or known contraindication to:

   1. Dipyridamole
   2. Ultrasound contrast agents (including PB127 and excipients)
   3. Blood, blood products, albumin, egg, or protein
3. Use of caffeine or xanthine containing products within the 24 hours prior to Study Day 1
4. Previous exposure to PB127 Ultrasound Contrast Agent
5. Major surgery within 7 days prior to Study Day 1 (requiring general anesthesia and/or overnight stay)
6. Heart transplant or history of CABG
7. Known hemodynamically significant or symptomatic right-to-left shunt (including shunts that are associated with prior TIAs or strokes)
8. Recent history of sustained ventricular tachycardia
9. Pacemaker or defibrillator
10. Unstable cardiac status

    1. Unstable angina grade CCS Class IV severity (any physical activity causes limiting symptoms; symptoms may be present at rest in a patient with prior exertional angina) with ongoing symptoms and/or ongoing infusion of intravenous nitroglycerin
    2. Decompensated heart failure
    3. Second-degree or greater heart block, sick sinus syndrome
    4. Frequent (>60/hour) or symptomatic ventricular ectopics at baseline
    5. Hypertension (SBP >200 and/or DBP >110 mmHg on two consecutive readings within one hour of PB127 MPE)
    6. Hypotension (SBP <90 mmHg)
    7. Severe aortic stenosis (>40 mmHg mean gradient or <0.6 cm2/m2 valve area index)
    8. Pulmonary edema within the 7 days prior to Study Day 1
    9. Resting oxygen saturation of less than 90% on room air
11. Myocardial infarction or cerebral vascular accident / transient ischemic attack within the 28 days prior to Study Day 1
12. Chronic Obstructive Pulmonary Disease (COPD) or bronchospastic airway disease, which in the opinion of the Investigator, is significant enough to contraindicate dipyridamole
13. Known history of severe pulmonary hypertension characterized by estimated pulmonary artery systolic pressure of >50 mmHg
14. Liver disease characterized by one or more of the following

    1. Current jaundice
    2. Elevated bilirubin > upper limit of normal
    3. Currently elevated hepatic enzymes > 2X upper limit of normal
    4. Current or previous hepatic viral infection (not including hepatitis A)
    5. Chronic hepatitis
15. Medical conditions or other circumstances that would significantly decrease the chances of obtaining reliable data or achieving the study objectives (i.e., drug dependence, psychiatric disorder, dementia, or associated illness); extenuating circumstances or medical conditions that make it unlikely that a patient can complete the clinical trial or follow up evaluations; or other reasons for expected poor compliance with the clinical investigator's instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of PB127 MPE for the detection and/or exclusion of significant obstructive coronary artery disease as defined by qualitative coronary angiography or qualifying clinical outcome | 72 hours, 6 months

SECONDARY OUTCOMES:
To compare the diagnostic performance of PB127 MPE to SPECT for the detection and/or exclusion of significant obstructive coronary artery disease. | 72 hours, 6 months
To assess the concordance of PB127 MPE with SPECT in the differentiation of defect type (fixed versus reversible) in patients with significant obstructive CAD. | 72 hours, 6 months
To evaluate the diagnostic performance characteristics of PB127 MPE for identifying the location of significant obstructive CAD as defined by quantitative coronary angiography | 72 hours
To assess the change in diagnostic certainty when PB127 MPE and relevant clinical information are combined over relevant clinical information alone. | 72 hours, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ehlgen, MD, PhD, Study Director — POINT Biomedical Corp
Locations (40):
- United States (40):
  - University of Arizona Saver Heart Clinic, Tucson, Arizona
  - Cardiovascular Associates of the Peninsula, Burlingame, California
  - Long Beach VA Medical Center Cardiology Division, Long Beach, California
  - Cedars Sinai Medical Center Division of Cardiology, Los Angeles, California
  - Sutter Roseville Medical Center, Roseville, California
  - University of California San Diego Division of Cardiology, San Diego, California
  - San Francisco VA Medical Center NCIRE, San Francisco, California
  - Connecticut Clinical Research, Bridgeport, Connecticut
  - Alfieri Cardiology, Newark, Delaware
  - Washington Hospital Center Cardiovascular Research Institute, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Midwest Cardiology Associates, Overland Park, Kansas
  - The Center for Cardiovascular Studies Kramer & Crouse Cardiology, Shawnee Mission, Kansas
  - Western Baptist Hospital The Heart Group, Paducah, Kentucky
  - Androscoggin Cardiovascular Associates, Auburn, Maine
  - Maine Cardiology Associates, South Portland, Maine
  - Brigham & Women's Hosptial, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Department of Cardiology, Rochester, Minnesota
  - Cardiovascular Consultants, Kansas City, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - St. Luke's Roosevelt Hospital Echocardiography Lab, New York, New York
  - Stonybrook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Cardiology Associates, High Point, North Carolina
  - The Cleveland Clinic Foundation Department of Cardiology, Cleveland, Ohio
  - Ohio State University College of Medicine and Public Health, Columbus, Ohio
  - University of Oklahoma Health Sciences Center VA Medical Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Seton Healthcare Network Brackenridge Hospital, Austin, Texas
  - Austin Heart, Austin, Texas
  - Consultants in Cardiology, Fort Worth, Texas
  - University of Texas Division of Cardiology, Galveston, Texas
  - Methodist DeBakery Heart Center Cardiovascular Imaging Institute, Houston, Texas
  - University of Texas Health Science Center Memorial Hermann Heart & Vascular Institute, Houston, Texas
  - Harborview Medical Center Department of Cardiology, Seattle, Washington
  - Heart Clinics Northwest, Spokane, Washington
  - Inland Cardiology, Spokane, Washington
  - Northwest Cardiovascular Research Institute Spokane Cardiology, Spokane, Washington